CLINICAL TRIAL: NCT05688163
Title: Effects of a Daily Cognition Training Programme on Cognitive Function, Emotional State, Frailty and Functionality in Older Adults Without Cognitive Impairment
Brief Title: Effects of a Daily Cognition Training in Older Adults Without Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Salamanca
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Functional Status; Cognitive Impairment; Occupational Therapy
Keywords: Functional Status; Cognition Therapy; Cognitive Impairment; Occupational therapy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional cognitive stimulation (Active Comparator): The control group will carry out the programme based on traditional cognitive stimulation. Individual cognitive skills such as attention, memory, executive functions, orientation, praxis, calculation, visual perception and reasoning will be trained. The materials and media used will be a cognitive stimulation notebook created for the study which includes cards in printed paper format to be completed by the participants.
  Interventions: Other: traditional cognitive stimulation
- programme based on everyday cognition (Experimental): The experimental group, on the other hand, will carry out a programme based on everyday cognition, i.e. the use of cognitive functions to solve real everyday problems that occur in our daily lives and that allow us to be autonomous in our homes, such as preparing food, taking care of the house, using transport, shopping, using the telephone, medication, financial management and access to information and current affairs. As material for use as for the traditional cognitive stimulation sessions, a training booklet on everyday cognition has been created which includes all the sessions mentioned above.
  Interventions: Other: programme based on everyday cognition

INTERVENTIONS:
Other: programme based on everyday cognition — Will carry out a programme based on everyday cognition, As material for use as for the traditional cognitive stimulation sessions, a training booklet on everyday cognition has been created which includes all the sessions mentioned above. Each day one of these tasks will be worked on.
  Arms: programme based on everyday cognition
Other: traditional cognitive stimulation — Individual cognitive skills such as attention, memory, executive functions, orientation, praxis, calculation, visual perception and reasoning will be trained. The materials and media used will be a cognitive stimulation notebook created for the study which includes cards in printed paper format to be completed by the participants.
  Arms: traditional cognitive stimulation

SUMMARY:
To evaluate the effectiveness of a daily cognition training programme versus a traditional cognitive stimulation programme in cognitively unimpaired older adults on cognitive function, emotional state, frailty and functionality.

DETAILED DESCRIPTION:
The present study aims to demonstrate the effectiveness of programmes that use everyday cognition for the assessment and intervention of healthy elderly people with the aim of maintaining or improving autonomy, compared to other programmes based on traditional cognitive stimulation, whose benefits do not generalise to significant improvements in everyday life. In addition, the investigators seek to relate how the presence of depression in older people impacts on everyday cognition, and therefore on the functionality of IADLs.

2. WORKING HYPOTHESIS AND MAIN OBJECTIVES TO BE ACHIEVED

1. WORKING HYPOTHESES

   * Alternative hypothesis (H1): Everyday cognition training programmes are more effective than traditional cognitive stimulation on cognitive function, emotional state, frailty and functionality in older adults without cognitive impairment.
   * Null hypothesis (Ho): Everyday cognition training programmes are not more effective than traditional cognitive stimulation on cognitive function, emotional state, frailty and functionality in older adults without cognitive impairment.

   In order to validate or disprove the main hypothesis, the following objectives have been developed:
2. OBJECTIVES:

i. MAIN OBJECTIVE: To evaluate the effectiveness of a daily cognition training programme versus a traditional cognitive stimulation programme in older adults without cognitive impairment, for cognitive function, emotional state, frailty and functionality.

ii. SPECIFIC OBJECTIVES:

* To compare the differences in the emotional state of older adults without cognitive impairment between the everyday cognition training programme and traditional cognitive stimulation.
* To contrast the differences in the cognitive function of older adults without cognitive impairment between the daily cognition training programme and traditional cognitive stimulation.
* To analyse the differences in the frailty index of older adults without cognitive impairment between the daily cognition training programme and traditional cognitive stimulation.
* To identify the differences in the functionality of older adults without cognitive impairment between the daily cognition training programme and traditional cognitive stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 60 years or older.
* Voluntarily sign the informed consent form about the project, authorising their participation.
* Carry out the initial assessment.
* Be admitted to the programme from the start of the programme.

Exclusion Criteria:

* No literacy skills or significant deficits in language comprehension.
* Institutionalised person.
* Have a clinical diagnosis of cognitive impairment.
* Participate in another cognitive stimulation programme during the intervention process.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Everyday cognition. | 35 minutes
  The Test for the Assessment of Everyday Cognition measures the ability of older people to solve everyday problems through performance tasks whose resolution depends on their cognitive capacity. The abilities tested are planning ability and cognitive flexibility, verbal working memory, reasoning, episodic memory, episodic memory and crystallised intelligence. The result is a direct estimation of the person's functional capacity by means of 12 real situations grouped into 6 areas: medication, administrative management, financial management, meal preparation, transport and shopping. The administration time is about 35 minutes.

SECONDARY OUTCOMES:
Cognitive function. | 10 minutes
  MONTREAL COGNITIVE ASSESSMENT TEST (MoCA test) Versión 8.3. :It is a cognitive assessment tool created to detect mild cognitive impairment (MCI). It evaluates executive functions, attention, abstraction, memory, language, visual-constructive abilities, calculation and orientation. It takes approximately 10 minutes to administer. The maximum score is 30 points, below 26 points being the cut-off for MCI (in developed countries).
Emotional state. | 10minutes
  Yesavage: It is a screening questionnaire for depression in people over 65 years of age. The 15-item version was selected for this study. It expresses the degree of satisfaction, quality of life and feelings. Of the 15 items, 10 indicate the presence of depression if answered positively, while the remaining 5 items answered negatively indicate depression. The administration time is 5 minutes. A score above 5 shows moderate depression and above 10 severe depression.
Instrumental activities of daily living | 5 minutes
  LAWTON AND BRODY SCALE: This is an assessment designed to evaluate autonomy in IADLs in the elderly population. It consists of eight items: use of the telephone, shopping, meal preparation, housekeeping, laundry, transport, medication management, use of transport and money. It takes 4 minutes to administer and is scored 0 or 1 for each item, making a total score of 8. At present, it is influenced by a gender bias as it is more sensitive to women than men (many of the activities have been performed only by women throughout history).
Functionality. | 15 minutes
  FUNCTIONAL INDEPENDENCE MEASURE (FIM): This is a tool created to measure the level of functionality and assistance given by the caregiver. It assesses the activities of daily living subdivided into two dimensions: the motor dimension; which assesses self-care (feeding, personal grooming, bathing, upper body dressing, lower body dressing, perineal grooming), sphincter control (bladder and bowel), transfers (to and from the chair or wheelchair, transfer in the bathroom, bath or shower) and locomotion (walking or moving around in a wheelchair, going up or down stairs). And cognitive; which assesses communication (comprehension, expression) and social knowledge (social interaction, problem solving and memory). Each of the 18 items has a maximum score of 7 and a minimum score of 1, making a total of 126.
Fragility. | 5 minutes
  FRAILTY SCALE: This is an assessment designed to quantitatively measure frailty in geriatric patients. It consists of 5 questions on real-life situations in which some frailty may affect quality of life. The maximum score is 5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo José Fernández Rodríguez, Salamanca, España, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available upon request by contacting the following e-mail address: edujfr@usal.es.
Supporting Information: Study Protocol
Time Frame: From the start of recruitment until two years after the end of recruitment.
Access Criteria: All data will be made available upon request by contacting the following e-mail address: edujfr@usal.es.

REFERENCES:
- [Derived] Saez-Gutierrez S, Fernandez-Rodriguez EJ, Sanchez-Gomez C, Garcia-Martin A, Barbero-Iglesias FJ, Sanchez Aguadero N. Study protocol for a randomized controlled trial: Effect of an everyday cognition training program on cognitive function, emotional state, frailty and functioning in older adults without cognitive impairment. PLoS One. 2024 Mar 29;19(3):e0300898. doi: 10.1371/journal.pone.0300898. eCollection 2024. PMID 38551981